CLINICAL TRIAL: NCT02653937
Title: The Effect of Shigyakusan Used for Irritable Bowel Syndrome and Medically Unexplained Physical Symptoms Diagnosed by Abdominal N Line Tenderness
Brief Title: The Effect of Shigyakusan Used for IBS and MUPS Diagnosed by Abdominal N Line Tenderness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nakatani Clinic (Other)
Collaborators: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Masaki Nakatani, MD, Ph.D. Researcher in Wakayama Medical University, Nakatani Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2015-06-19; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; MUPS; FSS; shigyakusan; Katsumi's points; Nakatani's N line
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kampo medicine (Experimental): 7.5g per day of Tsumura's shigyakusan ( Tsumura & Co ) was administered to each of 110 cases.
  Interventions: Drug: Tsumura's shigyakusan

INTERVENTIONS:
Drug: Tsumura's shigyakusan — Shigyakusan appears in the early 3rd Century. Four herbal crude medicines included are the following:
  Root of Bupleurum falcatum L Unripe fruit of Citrus aurantium Linne var. daidai Makino, Citrus aurantium Linne, or Citrus natsu-daidai Hayata (Rutaceae) Root of Paeonia lactiflora Pall Root and stolon of Glycyrrhiza uralensis Fisher or Glycyrrhiza glabra Linne
  Other Names: There is no other name other than Tsumura's shigyakusan.

SUMMARY:
Abstract

Background & Aims:

Abdominal N line tenderness for diagnosis and shigyakusan for treatment of irritable bowel syndrome ( IBS ) and medically unexplained physical symptoms ( MUPS ) were studied.

K1 is point of one quarters of distance from center of navel to right anterior superior iliac spine. K2 is one quarters of distance from center of navel to upside of the symphysis pubis. K3 is center of line from xiphoid process to navel. There are three relevant lines; K1-K3 line, K2-K3 line, and line of identical length to K1-K3 line originating from K2 and running parallel to K1-K3 line. Author collectively named these 'N line'. There was not the study under author's investigation that effects of shigyakusan and other medicines were compared. Author confirmed existence of mild IBS, for whose patients existing largely, various expensive examinations are spent.

Method:

The author put pressure on N line by deep palpitation and judged of abdominal N line tenderness positive or negative.

Shigyakusan, a Kampo medicine, was administered to each of N line positive patients, of IBS by Rome III, of no IBS by Rome III, and of MUPS. The change of symptoms of IBS and MUPS by shigyakusan was showed with an arrow by self-declaration.

Conclusions:

Shigyakusan was more effective for IBS than previous medicines. IBS was diagnosed by Rome III and N line tenderness and author confirmed the existence of mild IBS which was diagnosed by N line tenderness with help of RomeIII. MUPS showed N line tenderness though patients complained of no abdominal symptoms. Shigyakusan was very effective for IBS, mild IBS and MUPS.

DETAILED DESCRIPTION:
Background & Aims

The common cause of both IBS and MUPS is generally considered to be mental stress.

The late prof. Masaharu Katsumi at the Wakayama Medical University found two tender points "K1" and "K2" for IBS forty seven years ago. The author found another tender point "K3''. K1 is one quarters of the distance from the center of the navel to the right anterior superior iliac spine. K2 is one quarters of the distance from the center of the navel to the upside of the symphysis pubis. K3 is the center of the line from the xiphoid process to the navel. There are three relevant lines; the K1-K3 line, the K2-K3 line, and the line of identical length to the K1-K3 line originating from K2 and running parallel to the K1-K3 line. The author named these lines "N line" collectively.

The author considers as follows. K1 is the concentration point of nerves coming from the right colon, while K2 is the concentration point of nerves coming from the left colon, i.e. inferior mesenteric plexus. K3 corresponds to the superior mesenteric ganglion. The K1-K3 line corresponds to the root of mesentery. The K2-K3 line corresponds to the abdominal aortic plexus. The line originating from K2 and running parallel to the K1-K3 line is the line that transverses a number of nerves originating from jejunum or ileum, entering side by side into the root of mesentery and running to the superior mesenteric ganglion.

IBS is now diagnosed by the diagnostic criteria formed by symptoms. However, the author considers that medical sign of N line tenderness makes reliable diagnosis.

There was not the study under author's investigation that effects of shigyakusan and other medicines were compared. The author confirmed the existence of mild IBS which was diagnosed by N line tenderness with the help of Rome III, for whose patients existing largely, various expensive examinations and many hours are spent. MUPS showed N line tenderness though the patients complain of no abdominal symptoms.

Method

The author put pressure on the N line slowly by deep palpitation to check for tenderness of the region, comparing N line to the tenderness of the other parts of abdomen. He judged of abdominal N line tenderness positive or negative.

Shigyakusan, a Kampo medicine, was administered to each of N line positive patients, of IBS diagnosed by Rome III, of no IBS by Rome III, and of MUPS who have not abdominal symptoms of IBS in this study. The author enrolled 110 out-patients who were treated by shigyakusan at the Corporate Nakatani Clinic for two years from March 2013 to February 2015.

The author thinks that double blind study is the best way that shigyakusan is prescribed to placebo for clear endpoint discovered though it is very difficult to the psychiatric disorder as IBS. However, this time the author assessed the self-declaration of the symptom's change. The change of the symptom was showed with an arrow by self-declaration. An entry format was adopted by showing Table 1 to the patients. For example, ③→① shows the change of symptoms from ③ Significantly bad to ① Almost no symptoms in Table 1. The author used shigyakusan regardless of diarrhea or constipation.

Study of shigyakusan used for IBS:

The author tried to compare previous drugs to shigyakusan. 7.5g per day of Tsumura's shigyakusan ( Tsumura & Co ) was administered to each of 30 cases of IBS to whom Trimebutine maleate, Polycarbophil calcium and Oxapium iodide had been described, and was administered to each of 18 cases of new patients of IBS and 21 cases of existing patients first treated as IBS.(Table2) These patients were diagnosed as IBS by Rome III and abdominal N line tenderness, undermentioned in 'Regarding abdominal tenderness of N line' (Table 6).

Study of shigyakusan used for mild IBS

The patients of no IBS by Rome III and of abdominal N line tenderness positive were diagnosed as mild IBS for the reason in 'Regarding abdominal tenderness of N line' undermentioned (Table 6).

Shigyakusan was used for each of the patients with IBS who have mild to severe gastrointestinal symptoms without or with only few other bodily complaints or psychobehavioral features[26] :

7.5g per day of Tsumura' shigyakusan was administered to each of 14 cases of mild IBS(Table 3).

Study of shigyakusan used for MUPS:

MUPS are patients' unexplained & uncertain physical symptoms which are difficult for doctors to find the medical causes though MUPS do not imply that physical causes do not exist. However, MUPS in this study are physical symptoms other than IBS. When shigyakusan was effective for a patient suffered from both physical symptoms of MUPS and abdominal symptoms of IBS, the author adopted IBS.

7.5g per day of Tsumura' shigyakusan was administered to each of 27 MUPS patients who had doubt of psychiatric morbidity, for whom the author found no medical scientific cause(Table4).

Concerning N line when the cause of symptoms was clear

The possibility that the patients are diagnosed as MUPS becomes high if the patients have physical symptoms and show abdominal N line tenderness. When the cause of symptoms was clear without unaccountable or unexplained symptoms by having been examining, the author put pressure on N line by deep palpitation, and the author enumerated the thirty patients' conditions or diseases causing symptoms ( Table5 ).

ELIGIBILITY:
Inclusion Criteria:

* good constitution for shigyakusan

Exclusion Criteria:

* weak constitution for shigyakusan

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of participants who were suffered from IBS or MUPS, prescribed shigyakusan and improved. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Masaki Nakatani, M.D. Ph.D., Principal Investigator — Department of Gastroenterology, School of Medicine, Wakayama Medical Universiyy

REFERENCES:
- [Result] Hausteiner-Wiehle C, Henningsen P. Irritable bowel syndrome: relations with functional, mental, and somatoform disorders. World J Gastroenterol. 2014 May 28;20(20):6024-30. doi: 10.3748/wjg.v20.i20.6024. PMID 24876725
- [Result] Riedl A, Schmidtmann M, Stengel A, Goebel M, Wisser AS, Klapp BF, Monnikes H. Somatic comorbidities of irritable bowel syndrome: a systematic analysis. J Psychosom Res. 2008 Jun;64(6):573-82. doi: 10.1016/j.jpsychores.2008.02.021. Epub 2008 Apr 28. PMID 18501257
- See also: PMID 20233451 — http://www.ibsgroup.org/